CLINICAL TRIAL: NCT07297056
Title: The Effect of Mindfulness-Based Psychoeducation Programme on Mindfulness, Self-Compassion and Forgiveness Tendencies of Patients With Bipolar Disorder: A Randomised Controlled Trial
Brief Title: Mindfulness Psychoeducation for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ömer USLU (Other)
Responsible Party: Sponsor-Investigator, Ömer USLU, Dr. Ömer Uslu, PhD - Principal Investigator, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMER-RCT-2025-BAB
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder (BD); Mindfulness-Based Stress Reduction; Mindfulness Meditation
Keywords: Bipolar disorder, forgiveness, mindfulness, psychiatric nursing, self-compassion.
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the experimental group (mindfulness-based psychoeducation) or the control group with no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Psychoeducation (Experimental): Participants will receive an 8-session mindfulness-based psychoeducation program.
  Interventions: Other: Mindfulness-Based Psychoeducation Program; Other: routine care
- Control: Routine Care (No Intervention): Participants in this arm will receive Routine Care provided by the psychiatric outpatient clinic. Routine Care includes standard follow-up, medication management, and usual clinical monitoring. No additional psychoeducation or mindfulness-based intervention will be provided during the study period.

INTERVENTIONS:
Other: Mindfulness-Based Psychoeducation Program — A structured 8-session mindfulness-based psychoeducation program including mindfulness exercises, psychoeducation, breathing techniques and adherence-support strategies.
  Arms: Mindfulness-Based Psychoeducation
Other: routine care — Standard outpatient psychiatric care delivered by the clinic. No additional psychoeducation or mindfulness intervention is provided.
  Arms: Mindfulness-Based Psychoeducation

SUMMARY:
This randomized controlled experimental study investigates the effectiveness of a mindfulness-based psychoeducation program on mindfulness, self-compassion, and forgiveness among individuals diagnosed with bipolar disorder. Bipolar disorder is a chronic psychiatric condition characterized by fluctuations in mood, energy, and functional capacity, often accompanied by emotional dysregulation, impaired insight, and challenges in interpersonal relationships. Psychosocial interventions that cultivate emotional awareness and adaptive coping may support recovery and enhance long-term functioning.

In this study, 40 clinically stable patients with bipolar disorder were randomly assigned to either an experimental group (n=20) or a control group (n=20). The experimental group received a structured mindfulness-based psychoeducation program, while the control group received no additional intervention beyond usual care. Participants completed pre- and post-intervention assessments using a personal information form, the Mindfulness Scale, the Self-Compassion Scale-Short Form, and the Heartland Forgiveness Scale.

Findings demonstrated that individuals who participated in the mindfulness-based psychoeducation program showed significantly greater improvements in mindfulness, self-compassion, and forgiveness compared with the control group. These results suggest that integrating mindfulness-based psychoeducation into routine care may promote emotional resilience, enhance illness insight, support symptom management, and strengthen interpersonal functioning in individuals with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder is a chronic and recurrent psychiatric condition characterized by significant fluctuations in mood, energy levels, and functional capacity. Although pharmacological treatment remains the cornerstone of managing manic and depressive episodes, many individuals continue to experience residual symptoms, emotional dysregulation, heightened stress reactivity, and interpersonal difficulties even during periods of clinical stability. These challenges highlight the need for holistic approaches that address not only symptom reduction but also emotional regulation, self-awareness, and psychological well-being.

Mindfulness-based interventions have gained increasing attention as a complementary therapeutic approach for individuals living with bipolar disorder. Mindfulness practices cultivate the ability to observe internal experiences-thoughts, emotions, and bodily sensations-with openness, acceptance, and non-judgment. This enhanced awareness may reduce automatic emotional reactions, support early recognition of mood changes, and promote more adaptive coping strategies. By helping individuals respond rather than react to internal and external stressors, mindfulness may foster a sense of emotional balance and psychological resilience that is particularly valuable in bipolar disorder.

A key component closely linked to mindfulness is self-compassion, which involves treating oneself with kindness, understanding, and emotional warmth during times of difficulty or perceived inadequacy. Individuals with bipolar disorder often struggle with self-criticism, guilt, and negative self-appraisal stemming from the chronic and disruptive nature of the illness. Enhancing self-compassion may therefore help reduce emotional distress, facilitate more adaptive self-management, and strengthen long-term recovery-oriented functioning.

Forgiveness-toward oneself, others, and uncontrollable life circumstances-represents another important mechanism that may contribute to emotional healing in bipolar disorder. Difficulties associated with the illness may lead to strained relationships, unresolved emotional conflicts, or lingering feelings of resentment or self-blame. Developing forgiveness may promote emotional release, reduce psychological burden, and support healthier interpersonal dynamics.

The mindfulness-based psychoeducation program evaluated in this study integrates these components into a structured framework designed to enhance both emotional skills and illness-related insight. The program includes guided mindfulness practices such as breathing awareness and body scan exercises, psychoeducation modules that address symptom patterns and mood regulation, and reflective activities aimed at cultivating compassionate awareness and forgiveness. Through these combined elements, the intervention seeks to strengthen self-regulation capacities, promote acceptance-based coping, and improve psychosocial well-being in individuals with bipolar disorder.

By targeting mindfulness, self-compassion, and forgiveness simultaneously, the program offers a comprehensive approach to supporting emotional stability and personal recovery. This integrated model has the potential to enhance illness management, improve interpersonal functioning, and reduce the psychological burdens commonly experienced by individuals living with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder according to DSM-5 criteria
* Age between 18 and 65 years
* Clinically stable for at least the past 3 months
* Able to communicate, read, and understand Turkish
* Receiving outpatient psychiatric follow-up
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Presence of acute psychotic symptoms requiring immediate hospitalization
* Comorbid intellectual disability, neurological disorder, or severe cognitive impairment
* Substance or alcohol dependence within the last 6 months
* Participation in any mindfulness-based or psychoeducational program within the last year
* Severe visual or hearing impairment preventing participation
* Any condition judged by the clinician to contraindicate participation in group sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
Change in Mindfulness Level (Mindful Attention Awareness Scale) | Baseline and 8 weeks
  Mindfulness level was assessed using the Mindful Attention Awareness Scale (MAAS), a self-report questionnaire consisting of 15 items. Total scores range from 15 to 90, with higher scores indicating greater levels of mindfulness. The outcome measure represents the change in total MAAS score from baseline to post-intervention.

SECONDARY OUTCOMES:
Between-group Differences in Post-intervention Mindfulness and Treatment Adherence Scores | 8 weeks
  Between-group differences in post-intervention scores were evaluated using the Mindful Attention Awareness Scale (MAAS) and the Medication Adherence Rating Scale (MARS).
  Mindfulness was assessed with the MAAS, a 15-item self-report scale with total scores ranging from 15 to 90, where higher scores indicate greater mindfulness.
  Treatment adherence was assessed using the MARS, which consists of 10 items, with total scores ranging from 0 to 10, where higher scores indicate better medication adherence.
  The outcome measure represents the comparison of post-test total scores between the experimental and control groups at the end of the intervention.
Post-intervention Mindfulness and Treatment Adherence Scores Between Groups | 8 weeks
  Post-intervention differences between the experimental and control groups were evaluated using the following scales:
  Mindfulness: Assessed with the Mindful Attention Awareness Scale (MAAS), a 15-item self-report scale with total scores ranging from 15 to 90. Higher scores indicate greater mindfulness.
  Treatment Adherence: Assessed with the Medication Adherence Rating Scale (MARS), a 10-item self-report scale with total scores ranging from 0 to 10. Higher scores indicate better adherence to prescribed treatment.
  The outcome measure represents the comparison of post-test total scores between groups at the end of the 8-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Uslu, PhD, RN, Principal Investigator — Söke Fehime Faik Kocagöz Hospital
Locations (1):
- Söke Fehime Faik Kocagöz Hospital, Aydin, Söke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to ethical and institutional restrictions. The dataset includes sensitive health information from patients diagnosed with bipolar disorder, and the informed consent process did not include permission for public data sharing. Therefore, in accordance with privacy regulations and ethical committee requirements, IPD will not be made available to other researchers